CLINICAL TRIAL: NCT06119204
Title: Trial to Determine Safety And Efficacy of a Digital Low-Calorie Diet Programme (SAFE-LCD) for Insulin-treated Adults Living With Type 2 Diabetes
Brief Title: SAFE-LCD Trial, for Insulin-treated Adults Living With Type 2 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Oviva UK Ltd (Other)
Collaborators: Hull University Teaching Hospitals NHS Trust (Other Government); University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SAFE-LCD study (IRAS:321277)
Record Dates: First submitted 2023-10-11; First posted 2023-11-07 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes Treated With Insulin; Diet Habit
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: This study is a single centre, parallel-group, randomised controlled trial,
Masking Description: Due to the nature of the intervention, participants will not be blinded, thus they will be aware of the group allocation. However, the statistician will be blinded to participant allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Oviva ODR-I programme) (Experimental): The intervention arm will follow Oviva ODR-I programe: a 12-week TDR of approximately 850 calories per day through four TDR products daily, supported by the digital scales, CBG meters and link to the OVIVA app.
  Interventions: Other: Oviva programme
- Control (NHS 12 weeks programme) (Active Comparator): The control group will follow usual care, which will be the NHS 12-week digital weight-loss programme
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Oviva programme — Total diet replacement for insulin-treated patients
  Arms: Intervention (Oviva ODR-I programme)
Other: Usual care — NHS 12 week weight loss programme
  Arms: Control (NHS 12 weeks programme)

SUMMARY:
SAFE-LCD study is a randomised controlled trial aiming to develop and evaluate a safe, cost-effective, easily accessible, digital Low-Calorie Diet (LCD) programme for insulin-treated adults with Type 2 diabetes (T2D), a world-first innovation.

The study plans to enrol 72 participants who will be randomly allocated to either receive the intervention or will be provided with weight loss advice suitable for insulin-treated patients through accessing the NHS 12-week weight loss plan. The intervention arm will follow Oviva Diabetes Remission Insulin (ODR-I) programme which includes expert dietitian coaching, support of a Diabetes Nurse, the Oviva app (with a 12-month weight prediction chart), a Capilar Blood Glucose (CBG) meters (for enhanced safety in view of concerns re hypo- and hyper-glycaemia), and BodyTrace weight scales.

If successful, this project will provide game-changing evidence for the support of insulin-treated T2D patients and for NHS commissioning of the digital Low-Calorie programme driving patient benefits and cost-savings.

DETAILED DESCRIPTION:
Insulin treatment in Type 2 diabetes (T2D) patients is linked to poorer quality of life and and increased risk of complications due to disease progression.

This research study will be a randomised control trial (RCT) which is the highest quality form of medical evidence. It aims to develop and evaluate a safe, efficacious, cost-effective, easily accessible, digital Low-Calorie Diet (LCD) programme for insulin-treated adults with Type 2 diabetes (T2D), a world-first innovation.

The study plans to enrol 72 participants who will be randomly allocated to either receive the intervention or will be provided with weight loss advice through accessing the NHS 12-week weight loss plan.

The intervention will involve a 12-week Total Diet Replacement (TDR) diet of approximately 850 calories per day through four TDR products daily, followed by a 6-week food reintroduction period and weight maintenance support for 8 months. Care will be delivered fully remotely by Oviva's Diabetes Specialist Dietitians and Diabetes Specialist Nurse. Treatment aims are to achieve weight loss, improve diabetes control quality of life and decrease or in some cases discontinue insulin treatment.

The evaluation of ODR-I with independent clinical and health-economic evaluations will be undertaken by University College London and Insight Health Improvement and will be published in respected academic journals.

This groundbreaking research has the potential to achieve significant reductions in insulin use and to transform the lives of tens of thousands of people living with Type 2 diabetes. It will also save the NHS millions- if it is rolled out to just 62,000 patients a year, it will save more than £229 million a year in Type 2 Diabetes management costs across medications, monitoring, and hospital and General Practitioner(GP) usage.

ELIGIBILITY:
Inclusion Criteria:

* Registered with a GP practice within the confirmed NHS site - Humber and North Yorkshire
* Diagnosis of type 2 diabetes treated with insulin
* Age 18-70 years inclusive
* BMI ≥30kg/m² (adjusted to ≥27 kg/m² in ethnic minority groups)
* Upper body weight limit of 180kg (if using BodyTrace scales)
* Ability to speak, read and receive care in English language
* Access to the internet and a personal email address
* Access to and ability to use a smartphone
* Willing to test blood glucose up to 7 times a day (for up to 4 months) to ensure clinical safety.
* Participants capable to provide written informed consent and willing to comply with the trial protocol

Exclusion Criteria:

* C-peptide <200 pmol/L AND positive Glutamic Acid Decarboxylase(GAD) antibodies assessing for misdiagnosed Type 1 diabetes and risk of diabetic ketoacidosis.
* Type 1 diabetes mellitus, Mitochondrial diabetes, Maturity-Onset Diabetes of the Young (MODY) diabetes or diagnostic uncertainty (e.g. dual codes on patient record) Type 2 diabetes with history of diabetic ketoacidosis (DKA) or ketosis prone
* Clinically assessed hypoglycemia unawareness (via GOLD score (11, 12))
* Concomitant medication use clinically deemed to affect metabolic rate and body weight
* A major cardiovascular event within 6 months
* Severe angina, uncontrolled arrhythmia or known prolonged QT syndrome
* Warfarin or Rivaroxoban therapy
* Estimated glomerular filtration rate (eGFR) of less than 30 mL/min/1.73m²
* A condition precipitating fluid overload (e.g. New York Heart Association class III-IV congestive heart failure)
* Active liver disease (except non-alcoholic fatty liver disease (NAFLD)
* Active gallstone disease or known presence of gallstones
* Active cancer, receiving cancer treatment or received cancer treatment within past 24 months
* Known proliferative retinopathy that has not been treated
* Uncontrolled epilepsy
* Uncontrolled thyroid dysfunction
* Active or suspected peptic ulcer disease
* Gout
* History of bariatric surgery (previous band/balloon allowed if removed<12 months)
* Clinically diagnosed with an active eating disorder
* Clinically significant diagnosed/self-reported psychiatric disease that may interfere with study compliance
* Known or suspected alcohol or recreational drug misuse
* Milk allergy (Nualtra, TDR allergens)
* Soya allergy (Nualtra, TDR allergens)
* Vegan (Nualtra, animal derived Vit D)
* Pregnancy or planning pregnancy within study period
* Lactating
* Currently on a weight management programme or had in last 3 months or had over 5% weight loss in previous 6 months
* Current participation in other clinical intervention trials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-09-08 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Weight loss | at 12 months
  absolute: kg weight loss

SECONDARY OUTCOMES:
The number of participants reducing or ceasing insulin | at month 3, 6, 12 and 24
The number of participants reducing or ceasing other diabetes medications | at month 3, 6, 12 and 24
The number of participants reducing or ceasing cholesterol medications | at month 3, 6, 12 and 24
The number of participants reducing or ceasing blood pressure medications | at month 3, 6, 12 and 24
Hba1c (mmol/l) changes | at month 3, 6, 12 and 24
Diabetes remission rate | at months 3, 6, 12 and 24
  HbA1c below 6.5% (48 mmol/mol) and cessation of all diabetes medication for at least 3 months
Fasting and 2 hour postprandial/random glucose (mmol/L) | 1 year, throughout the study
  (measured via CBG meters)
Weight loss | at 3, 6 and 24 months
  relative: %, incl. the proportion of people achieving >5%, >10%, >15%, and >20% body weight loss
Cardiovascular disease risk score (QRisk) | at months 12 and 24
  Low Risk: A risk score of less than 10% means that there is less than a one in ten chance of developing cardiovascular disease in the next 10 years. Moderate Risk: A risk score of 10-20% means that there is between a one to two in ten chance of developing cardiovascular disease in the next 10 years. High Risk : A risk score of 20% equates to at least a two in ten chance of developing cardiovascular disease in the next 10 years.
Diabetes-related emotional distress (DDS17) | at month 6, 12 and 24
  The scale is used to measure emotional distress related to diabetes. It yields 4 sub-scales (Emotional burden, Regimen-related distress, Physician-related distress and Interpersonal distress). An overall distress score based on the average responses on the 1-6 scale (1"not a problem" to 6 "a very significant problem'') for all 17 items.
  A mean question score of 3 or higher (moderate distress) as a level of distress worthy of clinical attention.
Diabetes Stigma Assessment Scale Type 2 (DSAS-2) | at months 6, 12, and 24
  DSAS-2 is a valid and reliable self-report measure of diabetes-related stigma. It consists of three subscales: Treated Differently, Blame and Judgment, and Self-stigma. The score can be calculated for each subscale and in total. The higher the score the bigger the stigma.
EuroQol 5 Dimension 5 Level (EQ-5D) | at month 6, 12 and 24
  EQ5D is a self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Higher scores indicate more severe or frequent problems.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Thozhukat Sathyapalan, Principal Investigator — Hull University Teaching Hospital
Locations (1):
- Hull University Teaching Hospital NHS Trust, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided